CLINICAL TRIAL: NCT06884228
Title: Effects of Vibrating Mesh Nebulisation in Patients With COPD During Non-invasive Ventilation (VMN-NIV)
Acronym: VMN-NIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 348845
Record Dates: First submitted 2025-02-27; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Non-invasive Ventilation
Keywords: vibrating mesh nebuliser; jet nebuliser
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Pilot randomised crossover trial
Masking Description: VMN and JN are easily distinguishable due to both their visible and audible signatures. It is therefore not feasible to blind the patient to the delivered intervention. The mode of nebulisation will be known to both the investigator and participant, and the absence of masking is acknowledged to be a potential source of bias. Analysis of NRD and spirometry will be masked as an offline analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1st Vibrating mesh nebulisation and 2nd jet nebulisation (Experimental): Participants will receive a single dose of salbutamol whilst on NIV via vibrating mesh nebulisation on their first visit. After a minimum 48-hour washout period, they will receive the same dose of salbutamol via jet nebulisation while on NIV.
  Interventions: Device: Vibrating mesh nebulisation; Device: Jet nebuliser
- 1st Jet nebulisation and 2nd vibrating mesh nebulisation (Experimental): Participants will receive a single dose of salbutamol whilst on NIV via jet nebuliser on their first visit. After a minimum 48-hour washout period, they will receive the same dose of salbutamol via vibrating mesh nebuliser while on NIV.
  Interventions: Device: Vibrating mesh nebulisation; Device: Jet nebuliser

INTERVENTIONS:
Device: Vibrating mesh nebulisation — Vibrating mesh nebulisation (VMN) uses a mesh membrane that oscillates at high frequency (typically 128kHz) to produce a stream of drug-carrying droplets of pre-determined size to be inhaled
Device: Jet nebuliser — Jet nebulisers use the flow of a gas (air or oxygen) to draw medication up through a capillary tube to generate small particles to be inhaled.

SUMMARY:
Assessment of the effects of vibrating mesh nebulisation versus jet nebulisation on the electrical activity of the muscles involved in breathing (neural respiratory drive), breathing mechanics (respiratory impedance measured by forced oscillation technique), respiratory flow, heart rate and rhythm, spirometry and breathlessness symptoms in patients with chronic obstructive pulmonary disease who require non-invasive ventilation.

DETAILED DESCRIPTION:
Background Chronic obstructive pulmonary disease (COPD) remains a leading cause of morbidity and mortality in the United Kingdom. Acute exacerbations of COPD (AECOPD) frequently necessitate hospitalisation, with standard treatment comprising nebulised bronchodilators, antibiotics, and systemic corticosteroids. Approximately 20% of patients hospitalised with AECOPD require non-invasive ventilation (NIV) to manage decompensated hypercapnic respiratory failure, often necessitating concurrent administration of nebulised therapy.

Home NIV use is increasing among COPD patients to improve respiratory symptoms, quality of life, reduce hospitalisation frequency, and enhance survival. These patients may also require nebulised bronchodilator therapy during NIV, particularly when managing acute exacerbations not severe enough to warrant hospitalisation.

Currently, two nebulisation modalities are used as standard of care for patients on NIV:

Jet nebulisation (JN) - the conventional delivery method Vibrating mesh nebulisation (VMN) - a newer technology that utilises a mesh membrane oscillating at high frequency to produce drug-carrying droplets of predetermined size

VMN has been developed to optimise drug delivery in various patient populations, including those who are spontaneously breathing, receiving invasive mechanical ventilation, or on NIV. This technology is designed to enhance pulmonary drug deposition while minimising residual drug volume post-nebulisation.

Previous research has demonstrated that VMN achieves superior pulmonary drug deposition during NIV compared to JN in both healthy subjects and stable COPD patients. VMN has also been shown to produce greater improvements in forced expiratory volume in one second (FEV₁) among hospitalised patients. However, the comparative effects of these nebulisation methods on physiological parameters such as neural respiratory drive and respiratory system impedance during NIV in COPD patients with chronic respiratory failure remain unexplored.

Study Objective This pilot randomised crossover trial aims to compare the physiological effects of vibrating mesh versus jet nebulisation of salbutamol during NIV in patients with chronic respiratory failure due to COPD.

Methods Study Design A randomised crossover trial with participants receiving both interventions with a 48-hour washout period between treatments.

Participants We will recruit 12 patients with COPD currently receiving NIV under the care of the Lane Fox Unit. All participants will provide written informed consent prior to study procedures.

Procedures

Following consent, we will record baseline data including:

NIV settings Anthropometric measurements Arterial blood gas analysis Clinical observations

Participants will be randomised to receive salbutamol via either VMN or JN during NIV. We will measure the following parameters at multiple time points within one hour after nebulisation:

Neural respiratory drive via parasternal electromyography Spirometry Respiratory impedance (mechanics of breathing)

Participants will self-report breathlessness using both a numerical scale and a validated scale.

After a minimum of 48-hour washout period, participants will return to repeat the protocol with the alternative nebuliser type.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD receiving home non-invasive ventilation for chronic respiratory failure under the Lane Fox Respiratory Service at Guy's and St Thomas' NHS Foundation Trust
* Tolerating home non-invasive ventilation for at least 4 hours/24 hours
* Aged 18-80 years old
* Able to communicate symptom burden to the research team
* Able to give informed consent for participation in the study
* Clinical stability, with no acute exacerbations of COPD for 2 weeks prior to enrolment

Exclusion Criteria:

* Severe, non-respiratory organ dysfunction including, but not limited to:

  * Congestive cardiac failure
  * Significant cardiovascular disease
  * End-stage malignancy
  * End-stage renal failure
* Acute pulmonary pathology requiring emergency treatment including, but not limited to:

  * Pneumonia
  * Pneumothorax
  * Pulmonary embolism
* Severe cognitive impairment
* Psychosocial factors that would preclude completion of the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-21 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in neural respiratory drive | NRD assessed on both visits at baseline and 5, 15, 30 and 60 minutes after nebulisation
  Change in neural respiratory drive (NRD) 30 mins following vibrating mesh or jet nebulisation with a bronchodilator (2.5mg salbutamol) during NIV. This will be measured using surface second intercostal space parasternal muscle EMG. This reflects the load-capacity relationship of the respiratory system and will likely decrease with more effective bronchodilation and secretion clearance.

SECONDARY OUTCOMES:
Respiratory System impedence | Both visits at baseline, 5 and 60 minutes post nebulisation therapy.
  Change in respiratory system impedance 5 and 60 minutes after vibrating mesh or jet nebulisation therapy with 2.5mg salbutamol during NIV. Respiratory system impedance will be assessed using the forced oscillation technique (FOT).
  Change in the difference in within-breath respiratory reactance at 5Hz (ΔXrs,5Hz) 5 and 60 minutes after vibrating mesh or jet nebulisation therapy with 2.5mg salbutamol during NIV, as measured by FOT
Symptom of Breathlessness (numerical rating scale) | At baseline and at 5, 15, 30 and 60 minutes post nebulisation on both visits
  Breathlessness numerical rating scale: This will allow patients to report their dyspnoea and how it may change with treatment. The scale ranges from 0 to 10, where 0 indicates no breathing difficulty and 10 represents maximal breathing difficulty.
Symptom of Breathlessness (modified Borg Dyspnoea scale) | At baseline and at 5, 15, 30 and 60 minutes post nebulisation on both visits
  Patient perception of breathlessness will be assessed using the modified Borg dyspnoea scale (mBorg). The scale ranges from 0 to 10 (whole numbers plus 0.5), where - indicates no breathing difficulty and 10 represents maximal breathing difficulty.
Transcutaneous CO2 Monitoring | At baseline and for 60 minutes following nebulisation
  Continuous transcutaneous carbon dioxide levels will be measured
Spirometry - Forced expiratory volume in 1 second | At baseline and during 1 hour after administration of nebuliser on both visits
  Spirometry measurements of Forced expiratory volume in 1s second (FEV1)
Spirometry - Forced vital capacity | At baseline and during 1 hour after administration of nebuliser on both visits
  Spirometry measurements of Forced vital capacity (FVC)
Spirometry ratio - FEV1/FVC | At baseline and during 1 hour after administration of nebuliser on both visits
  Spirometry measurements used to calculate the ratio FEV1/FVC
Cardiac rate | At baseline and for 60 minutes following nebulisation
  Assessment of cardiac rate at baseline and following administration of salbutamol via VMN and JN.
Cardiac rhythm | At baseline and for 60 minutes following nebulisation
  Assessment of cardiac rate and rhythm at baseline and following administration of salbutamol via VMN and JN.
Respiratory flow | At baseline and for 60 minutes following nebulisation
  Assessment of respiratory flow via pneumotrach at baseline and following administration of salbutamol via VMN and JN

OTHER OUTCOMES:
Arterial blood gas | At baseline on first visit
  Allows assessment of the persistence and severity of the respiratory failure in addition to being a safety check.

CONTACTS AND LOCATIONS:
Overall Officials: Eui-Sik Suh, MBBS MChem(Oxon) PhD FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Lane Fox Unit, St Thomas' Hospital, Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson AC, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church AC, Creagh-Brown B, Dodd JW, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson CM, Sovani M, Thomas L; BTS Standards of Care Committee Member, British Thoracic Society/Intensive Care Society Acute Hypercapnic Respiratory Failure Guideline Development Group, On behalf of the British Thoracic Society Standards of Care Committee. BTS/ICS guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. Thorax. 2016 Apr;71 Suppl 2:ii1-35. doi: 10.1136/thoraxjnl-2015-208209. No abstract available. PMID 26976648
- [Background] Plant PK, Owen JL, Elliott MW. Early use of non-invasive ventilation for acute exacerbations of chronic obstructive pulmonary disease on general respiratory wards: a multicentre randomised controlled trial. Lancet. 2000 Jun 3;355(9219):1931-5. doi: 10.1016/s0140-6736(00)02323-0. PMID 10859037
- [Background] Brochard L. Non-invasive ventilation for acute exacerbations of COPD: a new standard of care. Thorax. 2000 Oct;55(10):817-8. doi: 10.1136/thorax.55.10.817. No abstract available. PMID 10992531